CLINICAL TRIAL: NCT05304936
Title: A Phase 1b/2 Study of HCW9218, a Bifunctional TGF-β Antagonist/IL-15 Protein Complex, for Advanced Pancreatic Cancer
Brief Title: HCW9218 for Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCWPAN102
Record Dates: First submitted 2022-03-11; First posted 2022-03-31 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Advanced Pancreatic Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HCW9218 (Experimental): Experimental Arm: HCW9218
  Interventions: Drug: HCW9218

INTERVENTIONS:
Drug: HCW9218 — Bifunctional TGF-β antagonist/IL-15 protein complex

SUMMARY:
This is a Phase 1b/2, open-label, multi-center, competitive enrollment and dose-escalation study of HCW9218 in patients with advanced/metastatic pancreatic cancer.

DETAILED DESCRIPTION:
The study involves a Phase 1b dose escalation portion with up to 30 patients to determine the MTD using a 3+3 dose escalation design and to designate a dose level for the Phase 2 expansion phase (RP2D).

The Phase 2 portion of the study will consist of an expansion cohort of up to 39 patients receiving HCW9218 monotherapy at the RP2D level. An additional independent Phase 2 cohort of patients receiving HCW9218 at the RP2D level in sequence with gemcitabine and nab-paclitaxel will also be considered.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed unresectable, advanced/metastatic disease pancreatic cancer that has progressed on standard first-line (or second- or later line) systemic therapy (excepting progression within 6 months of end of adjuvant systemic chemotherapy); or that can no longer be treated with first-line systemic therapy due to subject's intolerance.
2. For dose escalation phase (Phase 1b), distant metastatic disease or advanced disease and not a candidate for down staging to resection For expansion phase (Phase 2), distant metastatic disease only
3. Prior radiation is allowed if the index lesion(s) remains outside of the treatment field or has progressed since prior treatment. Radiation therapy must have been completed at least 4 weeks prior to the baseline scan.
4. Age > 18 years
5. A life expectancy of at least 12 weeks
6. Laboratory tests performed within 14 days of treatment start:

   1. Absolute neutrophil count (AGC/ANC) ≥ 1,500/μL (≥1.5 × 109/L)
   2. Platelets ≥ 100,000/μL (≥ 100 × 109/L) [Subjects may be transfused not more than 1 unit of platelets within 2 weeks to meet this requirement]
   3. Hemoglobin ≥ 9 g/dL (>90g/L) [Subjects may be transfused not more than 2 units of pRBCs within 2 weeks to meet this requirement]
   4. Calculated glomerular filtration rate (GFR)* >40 mL/min OR serum creatinine ≤ 1.5 × ULN
   5. Total bilirubin ≤ 2.0 × ULN or ≤ 3.0 × ULN for subjects with Gilbert's syndrome
   6. AST, ALT, ALP ≤ 2.5 × ULN or ≤ 5.0 × ULN if liver metastasis present *using the following Cockcroft & Gault equation to calculate the eGFR for this study.

   eGFR in mL/min = [(140-age in years) × (weight in kg) × F]/(serum creatinine in mg/dL × 72), where F =1 if male; and 0.85 for female.
7. Adequate pulmonary function with PFTs > 50% FEV1 if symptomatic or prior known impairment
8. Negative serum pregnancy test within 14 days of treatment start if female and of childbearing potential (non-childbearing is defined as greater than one year postmenopausal or surgically sterilized)
9. Female subjects of childbearing potential must adhere to using a medically accepted method of birth control prior to screening and agree to continue its use for at least 28 days after the last dose of HCW9218 or be surgically sterilized (e.g., hysterectomy or tubal ligation) and males must agree to use a barrier method of birth control and agree to continue its use for at least 28 days after the last dose of HCW9218
10. Provide signed informed consent and HIPAA authorization and agree to comply with all protocol-specified procedures and follow-up evaluations

Exclusion Criteria:

Subjects with ANY of the following criteria are excluded from participation in the study (to be verified by Sponsor prior to subject enrollment):

1. History of clinically significant vascular disease, including any of the following within 6 months prior to start of study treatment: MI or unstable angina, percutaneous coronary intervention, bypass grafting, ventricular arrhythmia requiring medication, stroke or transient ischemic attack, symptomatic peripheral arterial disease
2. Marked baseline prolongation of QT/QTc interval (e.g., demonstration of a QTc interval greater than or equal to 470 milliseconds by Fridericia's correction)
3. Subjects with untreated CNS metastases are excluded. Subjects are eligible if CNS metastases are treated and subjects are neurologically stable for at least 2 weeks prior to enrollment. In addition, subjects must be either off corticosteroids, or on a stable or decreasing dose of ≤ 10 mg daily prednisone (or equivalent)
4. Anti-cancer treatment including surgery, radiotherapy, chemotherapy, other immunotherapy, or investigational therapy within 14 days before treatment start
5. Other prior malignancy except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the subject is currently in complete remission, or any other cancer from which the subject has been disease-free for 3 years after surgical treatment
6. Known hypersensitivity or history of allergic reactions attributed to compounds of similar chemical or biologic composition to the agents used in the study
7. Prior therapy with TGF-β antagonist, IL-15 or analogs
8. Concurrent herbal or unconventional therapy (e.g., St. John's Wort)
9. Known autoimmune disease requiring active treatment. Subjects s with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of enrollment. Inhaled or topical steroids, and adrenal replacement steroid doses ≤ 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease
10. Active systemic infection requiring parenteral antibiotic therapy. All prior infections must have resolved following optimal therapy.
11. Prior organ allograft or allogeneic transplantation
12. Known HIV-positive or AIDS
13. Women who are pregnant or nursing
14. Any ongoing toxicity from prior anti-cancer treatment that, in the judgment of the Investigator, may interfere with study treatment. All toxicities attributed to prior anti-cancer therapy other than peripheral neuropathy, alopecia, and fatigue must resolve to grade 1 (NCI CTCAE v5.0) or baseline before administration of the study treatment
15. Psychiatric illness/social situations that would limit compliance with study requirements
16. Other illness or a medical issue that in the opinion of the Investigator would exclude the subject from participating in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
Occurrence of Adverse Events and Treatment-Related Adverse Events | 12 Months
  Evaluate the safety profile (as outlined by incidence of adverse events (AEs) based on CTCAE v5) of HCW9218 monotherapy in subjects with advanced/metastatic pancreatic cancer who have progressed on or are intolerant of standard first-line therapy
Determine the maximum tolerated dose (MTD) | 12 Months
  Determine the maximum tolerated dose (MTD) and designate the recommended Phase 2 dose level (RP2D) for Phase 2 study of HCW9218 in HCW9218-treated subjects

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 12 Months
  To evaluate objective response rate (ORR) per RECIST version 1.1
Progression-Free Survival (PFS) | 12 Months
  To assess the progression-free survival (PFS) per RECIST version 1.1
Overall Survival (OS) | 12 Months
  OS is defined as the time from first administration of study intervention to the date of death due to any cause.
Duration of Response | 12 Months
  Duration of response is the time from response to progression or death.

CONTACTS AND LOCATIONS:
Overall Officials: Paula Bradshaw, MSN, MBA, RN, Study Director — VP, Clinical Business Operations
Locations (5):
- United States (5):
  - HonorHealth, Scottsdale, Arizona
  - National Institute of Health/ National Cancer Institute, Bethesda, Maryland
  - Washington University in St. Louis, St Louis, Missouri
  - Cleveland Clinic, Cleveland, Ohio
  - Medical University of South Carolina, Charleston, South Carolina